CLINICAL TRIAL: NCT00685178
Title: Clinical Trial of Topiramate for Cocaine Addiction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01DA021808 (NIH); R01DA021808 (NIH)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Cocaine Dependence
Keywords: addiction; drug dependence; stimulant
MeSH Terms: conditions — Cocaine-Related Disorders; Behavior, Addictive; Substance-Related Disorders | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 topiramate + CR (Experimental): topiramate and contingency reinforcement for urine sample confirming cocaine abstinence
  Interventions: Drug: topiramate; Behavioral: Contingency Reinforcement
- 2 topiramate + NonCR (Experimental): Topiramate and random reinforcement irrespective of cocaine use
  Interventions: Drug: topiramate
- 4 Placebo + NonCR (Placebo Comparator)
  Interventions: Drug: placebo + NonCR
- 3 Placebo + CR (Active Comparator): Placebo and contingency reinforcement for urine sample confirming cocaine abstinence
  Interventions: Behavioral: Contingency Reinforcement

INTERVENTIONS:
Drug: topiramate — topiramate powder 0mg - 150 mg with lactate in blind capsules. Two capsules dispensed daily. One capsule ingested under supervision at the methadone window. One capsule to be ingested at home at bedtime. Participant is expected to return the empty blister pack on the following day.
  capsules are administered from week 4 through 25 of the trial
  Other Names: topamax®; CAS 97240-79-4
  Arms: 1 topiramate + CR; 2 topiramate + NonCR
Behavioral: Contingency Reinforcement — monetary reward for self-reported cocaine abstinence confirmed by urine toxicology results
  Other Names: contingency management
  Arms: 1 topiramate + CR; 3 Placebo + CR
Drug: placebo + NonCR — participant receives placebo capsules and monetary reinforcers by chance, irrespective of cocaine use or abstinence
  Arms: 4 Placebo + NonCR

SUMMARY:
This is an outpatient clinical trial of topiramate for addressing cocaine dependence and reduction of cocaine associated behaviors in opiate dependent drug users maintained on methadone treatment.

The study aims to answer whether topiramate

1. is safe and acceptable to methadone patients
2. reduces cocaine use
3. helps with collateral problems such as alcohol abuse, tobacco dependence, anxiety, PTSD and/or pain symptoms. The study will also evaluate topiramate effect on neuro-cognitive performance.

DETAILED DESCRIPTION:
This is an outpatient clinical trial of topiramate treatment for cocaine dependence and reduction of cocaine-associated HIV risk behavior. Topiramate is of high current interest in this regard, having been identified my National Institute on Drud Abuse (NIDA) leadership as among only a small number of tested candidates providing a "positive signal" and warranting further clinical investigation (Vocci, 2005). Topiramate is a marketed antiepileptic that enhances the GABAergic system and antagonizes the glutamatergic system, both new targets in the search for anti-cocaine treatments. A published pilot trial has supported topiramate's efficacy, and it is especially intriguing as potentially beneficial against other disorders prevalent among drug users, such as mood, anxiety, panic disorders, PTSD, pain and cognitive dysfunction, that may contribute to drug use. Design/Methods: This is phase II, double-blind randomized (stratified) 4 group, 2x2 design, evaluating topiramate versus placebo under each of two levels of cocaine-abstinence motivation -- cocaine-abstinence-contingent versus non-contingent voucher incentives. Conduct will be in a methadone maintenance context to ensure adequate retention and adherence, with participants dually dependent on opioids and cocaine. The target topiramate stabilization dose is 300 mg/day (150 mg b.i.d.), with one dose per day being observed at the clinic. The voucher-incentive manipulation provides valuable information about the role of motivation in modulating medication effects; it also provides a positive control condition to document the sensitivity of the study methods for detecting therapeutic benefit. Enrollment will be 300 patients ( 240 completers, 60/group). Participation will be up to 33 weeks - Baseline/Placebo-Run-in (5 weeks), Randomized Medication Treatment (20 weeks, induction, stable dosing, taper), Randomized Voucher Treatment (12 weeks, embedded in Medication period), and Therapeutic Disposition (up to 8 weeks). Data analysis focuses on the 8-week period of stable dosing and concurrent vouchers. The primary outcome variable is days abstinent from cocaine, as determined by a combination of self-report and objective confirmation by quantitative urinalysis toxicology of cocaine metabolite levels and application of the "Preston" rule for determining abstinence. Secondary outcome variables are measures of adverse behaviors and symptoms commonly co-occurring in cocaine abusers (alcohol abuse, tobacco use, depression, anxiety, PTSD, pain, neuro-cognitive and psychomotor performance dysfunction) that may contribute to drug use and/or detrimental effects. Significance: This randomized controlled clinical trial will provide valuable information about the actions and therapeutic effectiveness of the promising candidate anti-cocaine pharmacotherapy topiramate, and about the conditions, correlates, and modulators of any observed effectiveness. It will also provide valuable methodological information contributing to the continuing evolution of clinical trial methods for evaluating potential drug abuse treatment medications.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 55 years old
* active opioid and cocaine dependence
* seeking treatment for cocaine and opioid dependence
* eligible for methadone maintenance per state and federal regulations
* able and willing to provide a urine sample thrice a week
* willing to answer questionnaires on a weekly basis
* willing to provide breath samples for presence of alcohol thrice weekly
* fluent in the English language

Exclusion Criteria:

* allergy to sulfonamide drugs
* diabetes, respiratory insufficiency, renal tubular acidosis, renal insufficiency, heart failure, liver insufficiency, chronic diarrhea, other chronic diseases predisposing to a risk of acidosis
* history of nephrolithiasis
* HIV positive individuals who meet AIDS criteria by CDC criteria or are taking antiretroviral medications
* serious psychiatric illness (psychosis, dementia)
* glaucoma or family history of glaucoma
* prostate hyperplasia, shy bladder, irritable bladder, difficulty providing urine samples on demand
* female participants: being pregnant, lactating, or unwilling to use an effective method of contraception
* use of antiepileptic agents
* benzodiazepine dependence
* latex allergy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2007-02; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annie Umbricht, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Umbricht A, DeFulio A, Winstanley EL, Tompkins DA, Peirce J, Mintzer MZ, Strain EC, Bigelow GE. Topiramate for cocaine dependence during methadone maintenance treatment: a randomized controlled trial. Drug Alcohol Depend. 2014 Jul 1;140:92-100. doi: 10.1016/j.drugalcdep.2014.03.033. Epub 2014 Apr 16. PMID 24814607
- See also: Umbricht A∗, DeFulio A, Winstanley EL, Tompkins DA, Peirce J, Mintzer MZ, Strain EC, Bigelow GE (2014) Topiramate for cocaine dependence during methadone maintenance treatment: a randomized controlled trial Drug and Alcohol Dependence 140:92-100 — http://dx.doi.org/10.1016/j.drugalcdep.2014.03.033

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 250 volunteers were consented and admitted into the study; however 171 were randomized into the study. 79 volunteers were excluded due to a variety of reasons including failure to attend, adverse events (not study related), incarceration, failure to comply with study procedures, insufficient cocaine positive urines, and pregnancy
Groups:
- 1 Topiramate + CR: topiramate and contingency reinforcement for urine sample confirming cocaine abstinence
  topiramate: topiramate powder 0mg - 150 mg with lactate in blind capsules. Two capsules dispensed daily. One capsule ingested under supervision at the methadone window. One capsule to be ingested at home at bedtime. Participant is expected to return the empty blister pack on the following day.
  capsules are administered from week 4 through 25 of the trial
  Contingency Reinforcement: monetary reward for self-reported cocaine abstinence confirmed by urine toxicology results
- 2 Topiramate + NonCR: Topiramate and random reinforcement irrespective of cocaine use
  topiramate: topiramate powder 0mg - 150 mg with lactate in blind capsules. Two capsules dispensed daily. One capsule ingested under supervision at the methadone window. One capsule to be ingested at home at bedtime. Participant is expected to return the empty blister pack on the following day.
  capsules are administered from week 4 through 25 of the trial
Period: Overall Study
Arm/Group | 1 Topiramate + CR | 2 Topiramate + NonCR | 3 Placebo + CR | 4 Placebo + NonCR
Started | 40 | 45 | 39 | 47
Completed | 27 | 26 | 27 | 33
Not Completed | 13 | 19 | 12 | 14
Not completed — Adverse Event | 1 | 5 | 2 | 4
Not completed — missed 3 consecutive methadone clin days | 7 | 5 | 2 | 6
Not completed — voluntary study discharge | 4 | 5 | 1 | 1
Not completed — incarcerated | 1 | 3 | 7 | 0
Not completed — administrative (disciplinary) discharge | 0 | 1 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Topiramate + CR | 2 Topiramate + NonCR | 4 Placebo + NonCR | 3 Placebo + CR | Total
Number analyzed (Participants) | 40 | 45 | 39 | 47 | 171
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 45 | 39 | 47 | 171
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (7) | 41 (7) | 40 (8) | 42 (7) | 42 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 19 | 24 | 82
  Male | 23 | 23 | 20 | 23 | 89
Region of Enrollment [Number; unit: participants]
  United States | 40 | 45 | 39 | 47 | 171

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Cocaine Positive Urine Samples Per Treatment Condition
Description: Percentage of cocaine positive urine samples as measured by Preston new use rule (50% reduction in cocaine metabolites from previous urine)
Time Frame: Urine samples collected 3 times weekly from week 1 through 26
Population: This study utilized an Intent-to-Treat (ITT) analysis. The ITT analysis includes all volunteers who signed informed consent, were randomized into the study's treatment conditions, and took at least 1 dose of study medication.
Measure: Number; unit: percentage of positive urine samples
Arm/Group | 1 Topiramate + CR | 2 Topiramate + NonCR | 3 Placebo + CR | 4 Placebo + NonCR
Number analyzed (Participants) | 40 | 45 | 39 | 47
percentage of positive urine samples | 45.4 | 42.7 | 53.5 | 46.5
Statistical Analysis 1: Comparison: 1 Topiramate + CR vs 2 Topiramate + NonCR vs 3 Placebo + CR vs 4 Placebo + NonCR; Test type: Superiority; p = 0.531, Chi-squared — Using the proportion of negative urine samples obtained, the four groups were compared to determine whether there are any group differences in cocaine abstinence (as measured by negative urine samples); F-value for main effect of Condition = 2.210 — F-value for main effect of Drug Condition

2. Secondary Outcome: Voucher Earnings
Description: Voucher earnings used as a measurement of contigency management (CM) or operate conditioning. Volunteers were rewarded vouchers of escalating monetary value for cocaine abstinence, as indicated by a cocaine negative urine sample. The first cocaine negative urine earned a $2.50 voucher, and the value increased by $1.50 for each subsequent cocaine negative sample. Volunteers were awarded a bonus of $10.00 for every three consecutive cocaine negative urine samples. Urine samples were collected 3 times per week, and vouchers were attainable between Weeks 8 and 20.
  Contingency management as a measurement of operant conditioning in which positive reinforcement is applied (in this case vouchers of monetary value) and cocaine abstinence
Time Frame: 12 weeks (Weeks 8-20)
Measure: Mean (Standard Error); unit: Dollars
Arm/Group | 1 Topiramate + CR | 2 Topiramate + NonCR | 3 Placebo + CR | 4 Placebo + NonCR
Number analyzed (Participants) | 40 | 45 | 39 | 47
Dollars | 421.25 (79.58) | 343.26 (65.34) | 394.69 (72.06) | 203.51 (50.89)
Statistical Analysis 1: Comparison: 1 Topiramate + CR vs 2 Topiramate + NonCR vs 3 Placebo + CR vs 4 Placebo + NonCR; Analyses were performed to measure the correlation between CR groups (topiramate + CR and Placebo + CR) and abstinence; Test type: Superiority; p < 0.001, ANOVA; Spearmann's rank correlation = 0.969 — CR subjects only
Statistical Analysis 2: Comparison: 1 Topiramate + CR vs 2 Topiramate + NonCR vs 3 Placebo + CR vs 4 Placebo + NonCR; Analyses were performed to measure the correlation between Non-CR groups (topiramate + NonCR and Placebo + NonCR) and abstinence; Test type: Superiority; p < 0.001, Generalized Estimating Equation (GEE); Spearmann's rank correlation = 0.494 — NonCR subjects only

ADVERSE EVENTS:
Time Frame: 28 weeks (between Week 3 and Week 31)
Description: Standard Terminology.
  Reported adverse events include particpants who were randomized into the study's conditions (topiramate + CR/NonCR; placebo + CR/NonCR), and of which were rated as being either possibly, probably, or definitely related to the study.
Groups:
- 1 Topiramate + CR: topiramate and contingency reinforcement for urine sample confirming cocaine abstinence
  topiramate: topiramate powder 0mg - 150 mg with lactate in blind capsules. Two capsules dispensed daily. One capsule ingested under supervision at the methadone window. One capsule to be ingested at home at bedtime. Participant is expected to return the empty blister pack on the following day.
- 2 Topiramate + NonCR: Topiramate and random reinforcement irrespective of cocaine use
  topiramate: topiramate powder 0mg - 150 mg with lactate in blind capsules. Two capsules dispensed daily. One capsule ingested under supervision at the methadone window. One capsule to be ingested at home at bedtime. Participant is expected to return the empty blister pack on the following day.
Arm/Group | 1 Topiramate + CR | 2 Topiramate + NonCR | 3 Placebo + CR | 4 Placebo + NonCR
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/45 | 0/39 | 0/47
Serious Adverse Events (participants affected / at risk) | 4/40 | 4/45 | 1/39 | 3/47
Other Adverse Events (participants affected / at risk) | 1/40 | 5/45 | 3/39 | 3/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Topiramate + CR (N=40) | 2 Topiramate + NonCR (N=45) | 3 Placebo + CR (N=39) | 4 Placebo + NonCR (N=47)
Accidental CO Poisoning (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient Creatinine elevation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paranoid Psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases elevated (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased intraocular pressure (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pregnancy (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal EKG (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Topiramate + CR (N=40) | 2 Topiramate + NonCR (N=45) | 3 Placebo + CR (N=39) | 4 Placebo + NonCR (N=47)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (3) | 2 (2)
ECG Abnormal (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No